CLINICAL TRIAL: NCT02991196
Title: A Phase 1 Study of TRAIL-R2 (DR5) Antibody DS-8273a Administered in Combination With Nivolumab in Subjects With Advanced Colorectal Cancer
Brief Title: Antibody DS-8273a Administered in Combination With Nivolumab in Subjects With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DS8273-A-U103; Protocol ID CA209-860 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Neoplasm
Keywords: Advanced colorectal cancer; DNA mismatch repair (MMR); MMR-proficient Subjects; TRAIL-R2 (DR5) Antibody
MeSH Terms: conditions — Colorectal Neoplasms | interventions — DS-8273a; Nivolumab

ARMS (1):
- DS-8273a + nivolumab (Experimental): Participants will receive their treatment dose until discontinuation for any reason, or trial completion, within two years
  Interventions: Drug: DS-8273a + nivolumab

INTERVENTIONS:
Drug: DS-8273a + nivolumab — Nivolumab will be administered at 240 mg intravenously (IV) once every two weeks (Q2W) over 30 (± 5) minutes (on Days 1 and 15 of each cycle of 28 days). DS-8273a will be administered [90 (± 15) minutes on Day 1 of Cycle 1, and 60 (± 15) minutes in subsequent infusions] after the end of the nivolumab infusion in ascending doses up to 1200 mg IV Q2W. The regimen is adjusted based on injection site reactions or adverse events. Additional dose combinations may be considered based on the assessment of safety, primary pharmacodynamic (PDy) effects, and preliminary anti-tumor activities.

SUMMARY:
This trial is being performed in two parts: Dose Escalation and Dose Expansion.

The primary objective for the Dose Escalation part is to determine the safety and tolerability at different doses of DS-8273a administered in combination with nivolumab and to identify the dose combination for the Dose Expansion cohort in subjects with mismatch repair (MMR)-proficient advanced colorectal cancer.

The primary objectives for the Dose Expansion part are:

* To further evaluate the safety and tolerability of DS-8273a administered at the selected dose in combination with nivolumab in subjects with MMR-proficient advanced colorectal cancer
* To evaluate preliminary anti-tumor activity of DS-8273a plus nivolumab administered at the selected dose in subjects with MMR-proficient advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. A pathologically documented colorectal cancer that:
2. Is unresectable or metastatic
3. Has undergone ≥ 2 prior standard therapies
4. Is MMR-proficient [selected by the site based on microsatellite instability assay (MSI) and/or immunohistochemistry (IHC) for MMR proteins]
5. At least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
7. Peripheral blood MDSC level ≥ 10% of mononuclear cell fraction (assayed at a central laboratory)
8. Adequate bone marrow, renal, hepatic, and blood clotting function
9. Able to comply with protocol visits and procedures
10. Agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study (women for 23 weeks and men for 31 weeks after the last dose of study drug)
11. Are fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Institutional Review Board (IRB)-approved informed consent form (ICF), including Health Insurance Portability and Accountability Act authorization, if applicable, before performance of any study-specific procedures or tests
12. Are willing to provide available pre-existing diagnostic or resected tumor samples. Providing fresh tumor biopsies are optional for all subjects in Dose Escalation cohorts. In the Dose Expansion cohort, up to 6 subjects may be requested to provide pre- and post-treatment tumor biopsies based on eligibility for the procedure. For those subjects who do not have an MMR status, inclusion in the Dose Escalation and Dose Expansion can be achieved by providing a fresh tumor biopsy for MMR testing.
13. Subjects with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study. Inhaled steroids and intra-articular steroid injections are permitted in this study.

Exclusion Criteria:

1. Active infection or chronic comorbidity that would interfere with therapy
2. History of other malignancy(ies), except adequately treated non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥ 3 years.
3. History of severe hypersensitivity reactions to other monoclonal antibodies.
4. Any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that requires concomitant use of chronic systemic corticosteroids or other immunosuppressive medications, except for subjects with vitiligo, treated thyroiditis or resolved asthma/atopy.
5. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-cytotoxic T-lymphocyte-associated protein-4 (CTLA-4) antibody (or any other antibody targeting T-cell co-stimulation pathways).
6. Tested positive for hepatitis B or C serological markers (hepatitis B surface antigen or antibodies to hepatitis C virus) or human immunodeficiency virus.
7. Recipient of vaccines within 1 month of or during study drug treatment.
8. Requires daily supplemental oxygen.
9. Recipient of a stem cell or bone marrow transplant.
10. A concomitant medical condition that would increase the risk of toxicity, in the opinion of the Investigator or Sponsor.
11. Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.

    Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 4 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (2 weeks for stereotactic radiotherapy).
12. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. Subjects with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator after consultation with the Sponsor Medical Monitor or designee (eg, Grade 2 chemotherapy-induced neuropathy).
13. Systemic treatment with anticancer therapy, antibody-based therapy, retinoid therapy, or hormonal therapy within 3 weeks before study drug treatment; or treatment with nitrosoureas or mitomycin C within 6 weeks before study drug treatment; or treatment with small-molecule targeted agents within 2 weeks, or 5 half-lives before study drug treatment, whichever is longer.
14. Therapeutic radiation therapy or major surgery within 4 weeks before study drug treatment or palliative radiation therapy within 2 weeks before study drug treatment.
15. Participation in a therapeutic clinical study within 3 weeks before study drug treatment (for small-molecule targeted agents, this non-participation period is 2 weeks or 5 half-lives, whichever is longer), or current participation in other investigational procedures.
16. Pregnant or breastfeeding, or planning to become pregnant.
17. Substance abuse or medical conditions such as clinically significant cardiac or pulmonary diseases or psychological conditions, that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
18. Life expectancy < 3 months, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Part: Number of Participants with Dose-Limiting Toxicities (DLT) | During the first treatment cycle (28 days)
  A DLT is defined as a study drug-related ≥ Grade 3 Adverse Event (AE) occurring during the first cycle (28 days) of treatment, with specific exceptions for hematologic events, elevations in hepatic function enzymes, and adverse events that are pre-identified as not being DLTs.
Dose Escalation and Dose Expansion Parts: Number of Participants with Clinically Significant Safety Parameters | 2 years
  Safety parameters will include adverse events that are serious (SAEs), treatment emergent (TEAEs), dose-limiting toxicities (DLTs), physical examination findings (including Eastern Cooperative Oncology Group [ECOG] Performance Status), vital sign measurements, clinical laboratory parameters (serum chemistry, hematology, and urinalysis), immune-related (ir) adverse events (irAEs), anti-drug antibody (ADA), and electrocardiogram (ECG) parameters.
Dose Escalation Part: Maximum Tolerated Dose (MTD) | 2 years
  The MTD is defined as the highest dose of DS-8273a in combination with the tested dose of nivolumab that results in a DLT in less than one-third of the subjects enrolled at that dose level of at least 6 evaluable subjects. However, AEs that meet the definition of DLT appearing at later cycles will also be considered for the determination of MTD and selection of the Dose Expansion dose. If the MTD is not reached at 1200 mg of DS-8273a IV Q2W, this highest tested dose may be selected as the maximum administered dose (MAD).
Dose Expansion Part: Overall Objective Response Rate (per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1) | 2 years
  The overall objective response rate (ORR) is defined as the number of subjects whose Best Overall Response is either a Complete Response (CR) or Partial Response (PR), divided by the total number of treated subjects with at least one post-baseline tumor assessment.
Dose Expansion Part: Number of Participants in each Category of Best Overall Response (per Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1) | 2 years
  Categories: CR, PR, Stable Disease (SD), Progressive Disease (PD)
Dose Expansion Part: Disease Control Rate (DCR) for 6 Months | 6 months
  DCR for 6 months defined as the number of subjects with CR, PR, or SD for 6 months divided by the total number of treated subjects with at least 1 post-baseline tumor assessment
Dose Expansion Part: Number of Participants with Progression-Free Survival (PFS) | 2 years
  PFS is defined as survival without disease progression
Dose Expansion Part: Time to Progression (TTP) | within 2 years
  Mean TTP within 2 years
Dose Expansion Part: Duration of Response | within 2 years
  Duration of response for those subjects with a Best Overall Response of CR or PR
Dose Escalation Part: Number of Participants with Immune-related Response (per Criteria Modified from RECIST Version 1.1 [irRECIST]) | 2 years
  Criteria include:
  * Immune-related (ir) Best Overall Response with response categories of irCR, irPR, irSD, irPD
  * Immune-related ORR (irORR) defined as the number of subjects whose Best Overall Response is either an irCR or irPR divided by the total number of treated subjects with at least 1 post-baseline tumor assessment
  * Duration of immune-related-response for those subjects with immune-related Best Overall Response of irCR or irPR
  * Immune-related DCR (irDCR) for 6 months defined as the number of subjects with irCR, irPR, or irSD for 6 months divided by the total number of treated subjects with at least 1 post-baseline tumor assessment
  * Immune-related PFS
  * Immune-related TTP

SECONDARY OUTCOMES:
Plasma Concentrations of DS-8273a | Before and at the end of the first 3 infusions (Cycle 1 Days 1 and 15, and Cycle 2 Day 1), a single time point on Cycle 1 Day 8, then every 16 weeks on the same days as ADA sample analysis, and at the last Visit (if not collected within prior 16 weeks)
  The plasma concentrations of DS-8273a may be used to assess the exposure levels and for population pharmacokinetic (PK) analysis, if feasible, but no PK parameters will be calculated from the concentrations collected from this study due to sparse sampling time points.
Number of Participants with Primary Pharmacodynamic (PDy) Effects of the Combination Regimen on Myeloid-Derived Suppressor Cells (MDSCs) and their Subsets in Peripheral Blood | 2 years
  Subset Categories: Polymorphonuclear (PMN)-type and Monocytic-MDSCs (M-MDSCs)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Daiichi Sankyo
Locations (4):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/